CLINICAL TRIAL: NCT07031271
Title: Investigation of the Effect of Tangram Game on Patient Outcomes in Patients Undergoing Abdominal Surgery: A Randomised Controlled Study
Brief Title: The Effect of the Strategic Game Tangram on Postoperative Patient Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ezgi Arslan, PhD, Research Assisstant (Principal Investigator), Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Diversion of Attention
Record Dates: First submitted 2025-06-13; First posted 2025-06-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Pain Management; Postoperative Care; Nursing Care
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tangram game (Experimental): In this group, researchers will apply the Patient Identification Form to patients who are on the first day after surgery, who give at least 2 points for pain level, and who have had at least 3 hours since the last analgesic application, and will ask about the patients' pain and fatigue levels (First measurement). After this evaluation, patients in the intervention group will be asked to play the game for 20 minutes by making their own models with 7-piece tangram pieces in accordance with the randomization output. After the game, the pain and fatigue levels will be questioned again (Second measurement). The pain and fatigue levels will be questioned again 30 minutes after the second measurement (Third measurement).
  Interventions: Behavioral: Tangram game
- Usual care (No Intervention): In this group, researchers will apply the Patient Identification Form to patients who are on the first day after surgery, who give at least 2 points for pain level, and who have had at least 3 hours since the last analgesic application, and will ask about the patients' pain and fatigue levels (First measurement). After this assessment, no intervention will be applied to the patients, and the pain and fatigue levels will be questioned again 20 minutes after the first measurement (Second measurement). The pain and fatigue levels will be questioned again 30 minutes after the second measurement (Third measurement).

INTERVENTIONS:
Behavioral: Tangram game — Tangram game; It is a very old intelligence and attention game of Chinese origin. This game stands out with its both entertaining and educational aspects. Tangram consists of seven geometric pieces formed from a square shape. These 7 pieces; 2 large right triangles, 1 medium right triangle, 2 small right triangles, 1 square and 1 parallelogram. The aim is to create various shapes (animals, people, objects, letters, etc.) with these pieces. The aim of the Tangram game is to recreate the same appearance with a given shape (silhouette) using the pieces. All 7 pieces must be used in the game, the pieces must not be overlapped, the pieces must not be cut or divided, the pieces can be rotated or turned according to the selected shape. For example, the person is asked to create a cat figure with these 7 pieces in accordance with the rules. This game is one of the non-pharmacological pain management techniques by diverting the attention of the patients. It is easy to apply and cheap.
  Arms: Tangram game

SUMMARY:
The aim of this study was to investigate the effects of playing tangram game after surgery on pain, fatigue and comfort levels in patients undergoing abdominal surgery.

DETAILED DESCRIPTION:
Tangram game is a skill and strategy game based on creating 100 different forms, made of 4 or 7 pieces, made of wood. 100 different shapes are obtained by using all the given pieces. These patterns should be arranged from easy to difficult by following a given guide. Tangram game is a strong stimulant as it appeals to both visual and mental skills. Strong stimulants prevent the ongoing pain stimulus at that moment. Pain transmission is interrupted and the individual is prevented from feeling pain. During and after the game, the pain level begins to decrease thanks to different stimulants. Applications that give the individual pleasure, such as Tangram, provide the secretion of substances such as enkephalin and endorphin. With these secreted substances, the body's own analgesia system is supported and the severity of pain is reduced. There are studies in the literature testing non-pharmacological interventions in the management of post-operative pain and fatigue. Some of these studies include studies evaluating the effects of massage, listening to music, cold application, distraction strategies such as playing a tangram game or giving auditory stimulation, mobilization, reflexology, chewing gum, and acupuncture. There are limited studies in the literature on the use of tangram games in the management of postoperative pain, and no studies have been found examining the effects of this intervention on pain, fatigue, and patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Having had abdominal surgery
* Being on the first day after surgery
* Having a first pain measurement score of at least 2
* Having at least 3 hours since the last analgesic application

Exclusion Criteria:

* Having hearing/vision/mental problems
* Having limited movement in the hand/wrist/arm
* Having undergone surgery due to cancer
* Being diagnosed with a psychological illness (schizophrenia, depression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Pain level | Postoperative 1st day
  The numerical rating scale to be used in the assessment of pain is a one-dimensional 10 cm scale based on the patient's self-report. The lower end is "no pain", corresponding to 0 points, and the upper end is "unbearable pain", corresponding to 10 points. As the pain intensity expressed by the patient increases on the scale, it will be interpreted that the patient's pain increases. This is first measurement.
Pain level | 20 minutes later after first measurement
  The numerical rating scale to be used in the assessment of pain is a one-dimensional 10 cm scale based on the patient's self-report. The lower end is "no pain", corresponding to 0 points, and the upper end is "unbearable pain", corresponding to 10 points. As the pain intensity expressed by the patient increases on the scale, it will be interpreted that the patient's pain increases. This is second measurement.
Pain level | 30 minutes later after second measurement
  The numerical rating scale to be used in the assessment of pain is a one-dimensional 10 cm scale based on the patient's self-report. The lower end is "no pain", corresponding to 0 points, and the upper end is "unbearable pain", corresponding to 10 points. As the pain intensity expressed by the patient increases on the scale, it will be interpreted that the patient's pain increases. This is third measurement.
Fatigue level | Postoperative 1st day
  The numerical rating scale to be used in the assessment of fatigue is a one-dimensional 10 cm scale based on the patient's self-report. The lower end is "not tired" corresponding to 0 points, and the upper end is "unbearably tired" corresponding to 10 points. As the fatigue intensity expressed by the patient increases on the scale, it will be interpreted as the patient's fatigue increasing. This is first mesurement.
Fatigue level | 20 minutes later after fist measurement
  The numerical rating scale to be used in the assessment of fatigue is a one-dimensional 10 cm scale based on the patient's self-report. The lower end is "not tired" corresponding to 0 points, and the upper end is "unbearably tired" corresponding to 10 points. As the fatigue intensity expressed by the patient increases on the scale, it will be interpreted as the patient's fatigue increasing. This is second mesurement.
Fatigue level | 30 minutes later after second measurement
  The numerical rating scale to be used in the assessment of fatigue is a one-dimensional 10 cm scale based on the patient's self-report. The lower end is "not tired" corresponding to 0 points, and the upper end is "unbearably tired" corresponding to 10 points. As the fatigue intensity expressed by the patient increases on the scale, it will be interpreted as the patient's fatigue increasing. This is third mesurement.

SECONDARY OUTCOMES:
Comfort level | 30 minutes after second measurement
  General Comfort Scale-Short Form will be used to evaluate the comfort level. The scale consists of 28 items and the items of the scale are scored between 28-168. General Comfort Scale Short Form consists of three sub-dimensions: relief, relaxation, and superiority. GKÖ-SF was developed by Kolcaba in 2006 and its Turkish validity and reliability study was conducted by Çıtlık et al. in 2018. It includes the sub-dimensions of comfort, relief (9 items), relaxation (9 items), and overcoming problems (10 items). In the evaluation of the scale consisting of positive and negative items, the negative items are reverse coded and summed. The mean value is found by dividing the total score by the number of scale items. The lowest possible value, 1, indicates low comfort, and the highest value, 6, indicates high comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Aydin, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 12 months after publication
Access Criteria: Relevance to the topic of the study and approval of all-authors within 1 month of receiving the request.